CLINICAL TRIAL: NCT05389800
Title: Pre- and Post-Operative Effects of Upper Extremity Aerobic Exercise in Mobility, Haemostatic Balance, and Mortality- and Morbidity-related Biomarkers in Hip Fracture Patients: A Randomized Controlled Trial
Brief Title: Pre- and Post-Operative Exercise in Patients With Hip Fracture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Panagiotis Koulouvaris, MD, Assistant Professor, 1st Department of Orthopaedic Surgery, National and Kapodistrian University of Athens, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 402/26-7-2021
Record Dates: First submitted 2021-10-08; First posted 2022-05-25 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Hip Fractures
Keywords: hip fracture; exercise therapy; surgical stress; haemostasis; basic mobility
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Moderate-Intensity Interval Training) (Experimental): Preoperative program: 120 seconds of moderate intensity exercise (64-76% HRmax, 12-13 in rate of perceived exertion (RPE), based on ACSM) and 120 seconds of passive rest in a total of 4 cycles. The basic program will last about 14 minutes, plus 6 minutes for warm-up and recovery. The program will be performed twice a day.
  Postoperative program: 120 seconds of moderate intensity exercise (64-76% HRmax, 12-13 in RPE, based on ACSM) and 120 seconds of passive rest in a total of 8 cycles. The basic program will last about 30 minutes, plus 6 minutes for warm-up and recovery. The program will be performed 3 times a week for a total of 8 weeks.
  Interventions: Other: Upper Extremity Aerobic Exercise
- Control (No Intervention): Preoperatively: mild intensity activities focusing on memory and attention performing with upper limb movements using the interactive platform Kinems. The program will last about 20 minutes. To ensure that the intensity of activities is mild, there will be a simultaneous recording of heart rate, while at the end of each session the RPE scale will be evaluated.
  Postoperatively: none

INTERVENTIONS:
Other: Upper Extremity Aerobic Exercise — Using a cycle-ergometer (Monark 881E)
  Arms: Aerobic Exercise (Moderate-Intensity Interval Training)

SUMMARY:
The purposes of this study are to determine the benefits of a pre-operative aerobic exercise program and an 8-week postoperative aerobic exercise program with a portable upper extremity cycle-ergometer in patients with hip fracture.

DETAILED DESCRIPTION:
Hip fracture is one of the primary causes of significant morbidity in those over than 65 years old. Hip fracture is also among the top ten causes of loss of disability-adjusted life years in elderly. For the year 2020, in terms of the percentage of population over 80 years, Greece was second among the countries of the European Union, with this age group constituting 7.2% of its total population. In Greece, between 1977 and 2007, hip fractures doubled, with the annual impact rising to 343.96 per 100,000 inhabitants. For this population, a critical part of management is physical activity and exercise prescription both to prevent complications and to enhance rehabilitation after surgery. Postoperative (post-discharge) aerobic exercise programs of moderate intensity have already been used in patients with hip fracture proving its safety and positive effect in a variety of outcomes, such as aerobic capacity and quality of life. It is well established that these patients do not meet the minimum least amount of activity that should be done per week, based on Guidelines for Physical Activity by the World Health Organization neither during their hospitalization nor during their later life in the community. Also, although most Clinical Guidelines recommend a surgical management within 48 hours after hip trauma, there are many patient and system factors which can contribute to delayed surgery, such as surgical readiness, available resources, prioritisation and out-of-hours admission.

In terms of pre-operative exercise program, the investigators hypothesize that it will reduce surgical stress through the body's better response to lactate accumulation and the acute physiological effects on the patient's hematopoietic activity and hemostatic profile. Moderate intensity exercise will reduce platelet hyperactivity, increase fibrinolytic activity and reduce coagulation factors. In this more favorable environment, the immediate postoperative recovery of basic mobility can be accelerated. Regarding the post-operative exercise program, the investigators hypothesize that it will improve the independence and function of the lower extremity by increasing the cardiopulmonary capacity, while the improvement of the nutritional factors (albumin and pre-albumin) through the post-training protein synthesis will also contribute to this.

Apart from primary and secondary outcomes, at baseline the investigators will also evaluate the following: demographics; characteristics about the fracture and upcoming surgery, such as the type of fracture and the surgical procedure; New Mobility Score (NMS) to define the prefracture functional level; Addenbrooke's Cognitive Examination - III (ACE-III) to define the cognitive status.

The power analysis for the selection of the sample size for the postoperative program in the change of the 6-Minute Walk Test (primary outcome) after the completion of the program, in the 8 weeks postoperatively, was performed for significance level α = 0.05 and power = 90%.The investigators' assumption for power analysis stands to find a difference of 50 meters between the groups. Considering that the ratio between the groups will be 1: 1, the required sample size is 96 patients (48 in each group). Adding a drop-out rate of 20%, required sample size is defined in 116 patients (58 in each group). About the other primary outcome (postoperative 3-day Cumulated Ambulation Score - CAS), the investigators' power analysis revealed a required sample size of 80 patients, based on the assumptions of 2.4 points difference between the groups, α = 0.05 and power = 90%. In statistical analysis, only patients who completed at least a 3 days of preoperative program will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65 years old and older
* Unilateral proximal femoral fracture/hip fracture (intertrochanteric or neck fracture)
* Ambulatory patients before fracture (with or without aid assistance)
* Agreed to participate and signed consent form

Exclusion Criteria:

* Pathological fractures (under musculoskeletal oncology)
* Severe neuropsychiatric disorder (eg severe psychiatric disorder, dementia, etc.) to the extent that the researcher deems the patient incompetent or likely unable to remain compliant with the follow-up
* Unable to implement the exercise program due to underlying pathology or disability in the upper extremities
* More than one fracture
* Severe and / or unstable cardiovascular disease [e.g. congenital heart disease, uncontrolled severe hypertension (systolic blood pressure ≥ 180 mmHg and / or diastolic blood pressure ≥ 120 mmHg), unstable angina]
* Neurological or other conditions that significantly impair function and independence (eg stage 3-5 Parkinson's disease according to Hoehn and Yahr, advanced Multiple Sclerosis, severe arthritis of degenerative or rheumatic etiology)
* Severe metabolic bone disease (eg Paget's disease, renal bone disease, osteomalacia), excluding osteoporosis
* Active deadly aggressive disease (eg end-stage cancer with an estimated survival expectancy of less than 6 months)
* Unable to understand the consent document and / or protocol instructions
* Refusal to participate in the research

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cumulated Ambulation Score | Total 3-day Cumulated Ambulation Score post-operatively.
  The Cumulated Ambulation Score (CAS) is a reliable and valid instrument for assessing patients' basic mobility (getting in and out of bed, sit-to-stand from a chair, and walking), in orthopaedic wards. The minimum value is 0 and maximum 3 per day. The total 3-day CAS has a better prognostic value than the 1-day CAS, and is based on the sum score of the first three post-operative days, with a minimum value being 0 and maximum 9, for the total 3-day CAS, with a higher score means better outcome.
Six Minute Walk Test (6MWT) | 8 weeks post-operatively
  The 6MWT is a sub-maximal exercise test that is used to determine aerobic capacity and endurance.

SECONDARY OUTCOMES:
Cumulated Ambulation Score | 4 weeks post-operatively
  The Cumulated Ambulation Score (CAS) is a reliable and valid instrument for assessing patients' basic mobility (getting in and out of bed, sit-to-stand from a chair, and walking), in orthopaedic wards. Higher score means a better outcome.
Six Minute Walk Test (6MWT) | 4, 26 & 52 weeks post-operatively
  The 6MWT is a sub-maximal exercise test that is used to determine aerobic capacity and endurance.
Timed-Up & Go | 4, 8, 26 & 52 weeks post-operatively
  The Timed Up and Go (TUG) test is a performance-based measure of functional mobility that assess mobility and balance impairments in older adults. Patients wear their usual shoes and, if necessary, can utilize a walking assistance. Begin by having the patient sit back in a normal armchair and drawing a line on the floor 3 meters (10 feet) away.
Modified Harris Hip Score | At admission (for pre-operative status) and 4, 8, 26 & 52 weeks post-operatively (for current status)
  The modified Harris Hip Score (mHHS) is a reliable and valid self-reported questionnaire assessing hip pain and functionality. One question evaluates pain (score from 0-44) and 7 questions functionality (score from 0-47). The overall score is multiplied by 1.1 leading to a possible score of 0 to 100, with 100 being the best possible score for hip pain and function.
Lower Extremity Functional Scale | At admission (for pre-operative status) and 4, 8, 26 & 52 weeks post-operatively (for current status)
  The Lower Extremtiy Functional Scale (LEFS) is a reliable and valid self-reported questionnaire assessing lower extremity function. The LEFS consists of 20 questions, evaluated on a 5-point scale (0-4˙ 0 = extremely high degree of difficulty, 4 = no difficulty, with a total score up to 80 degrees).
Lactate levels | Day 0 (at admission), Intraoperatively (at the beginning, 30 minutes later, and at the end of the surgery), & 12h postoperatively
  Capillary blood with Lactate Scout+
Albumin levels | First day of admission, one day before surgery, 3 days, 4, 8, 26 & 52 weeks post-operatively
Tissue plasminogen activator | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
Plasminogen activator inhibitor-1 | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
Thrombin-Antithrombin Complex | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
Endogenous Thrombin Potential | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
Fibrinogen plasma levels | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
  The fibrinogen normal range is 200 to 400 mg/dL (2.0 to 4.0 g/L). Determination of fibrinogen plasma concentrations will be made performing a modification of the Clauss method with Fibrinogen Multifibren U reagent (Siemens Healthcare Diagnostics, Marburg, Germany). Fibrinogen increased levels are significantly associated with inflammatory markers, disease severity and thrombotic tendency.
  The effect of the pre-operative and post-operative aerobic exercise on this variable and its association with clinical outcome will be assessed.
D-Dimers plasma levels | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
  The reference concentration of D-dimer is < 250 ng/mL. D-dimers were assessed by the INNOVANCE D-Dimer assay (Siemens Healthcare Diagnostics, Marburg, Germany), a particle-enhanced immunoturbidimetric method. Besides the value of normal D-dimer measurements in allowing exclusion of venous thromboembolism (VTE) or pulmonary embolism (PE), D-dimer test also helps clinicians to stratify patients with the risk for deep venous thrombosis (DVT), since high levels of D-dimer in blood are associated with a major clot. That's why increased D-Dimer levels are considered as a marker of hemostatic imbalance.
  The effect of the pre-operative aerobic and post-operative exercise on this variable and its association with clinical outcome will be assessed.
Thrombomodulin plasma levels | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
  Thrombomodulin (TM)levels range from 3 to 300 ng/ml. with normal levels fluctuating between 3.1 ± 1.3 ng/ml. A TM sandwich ELISA double antibody kit will be used for the measurements. TM, which is predominantly expressed on the endothelium, plays an important role in maintaining vascular homeostasis by regulating the coagulation system. During the hypercoagulable state after endothelial injury, TM is released into the intravascular space, thus reflecting derangements of hemostatic balance due to endothelial dysfunction. Moreover, TM reduces blood coagulation by converting thrombin to an anticoagulant enzyme from a procoagulant enzyme, while it has the potential to regulate intravascular injury via pleiotropic effects.
  The effect of the pre-operative and post-operative aerobic exercise on this variable and its association with clinical outcome will be assessed.
von Willebrand factor (VWF); VWF:Antigen and VWF:Activity plasma levels | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
  VWF:Antigen(Ag) and VWF:Activity(Ac) are used as markers of Platelet and Endothelial Dysfunction affecting hemostatic balance. VWF:Ag and VWF:Ac plasma levels will be determined by an automated latex enhanced immunoassay (HaemosIL™ assay, Instrumentation Laboratory Company, Lexington, KY, USA) on IL (Instrumentation Laboratory) coagulation systems (ACL TOP). VWF:Ac will be assessed by measuring the variations in turbidity generated by the agglutination of the latex reagent. An anti-VWF monoclonal antibody adsorbed onto the latex reagent reacts with the VWF of the blood sample. Agglutination is proportional to VWF:Ac and is calculated by the diminished light transmission caused by the aggregates. Results are presented as percentage of normality.
  The effect of the pre-operative and post-operative aerobic exercise on this variable and its association with clinical outcome will be assessed.
Haemostatic profile using ROTEM | First day of admission, one day before surgery, 3 days, 1, 4, 8, 26 & 52 weeks post-operatively
Transfusion requirements (litre) | Post-operative day 1, 2 and 3
Deep vein thrombosis & Pulmonary embolism (DVT & PE) | 4, 8, 26 & 52 weeks post-operatively
  Number of every thromboembolic event
Re-admission | 4, 8, 26 & 52 weeks post-operatively
  Re-admission rate for any reason
All-cause mortality | 4, 8, 26 & 52 weeks post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Koulouvaris, MD, Principal Investigator — 1st Department of Orthopaedic Surgery, National and Kapodistrian University of Athens
Locations (1):
- 1st Department of Orthopaedic Surgery, Medical School, National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
The data of this study will be available from the corresponding author, upon reasonable request.